CLINICAL TRIAL: NCT00758316
Title: A Prospective, Randomized Controlled Trial for a Rapid Pleurodesis Protocol for the Management of Pleural Effusions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 149/2008
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Malignant Pleural Effusions
Keywords: Malignant; Pleural; Effusions; Thoracoscopy; Catheter
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Thoracoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Thoracoscopy with pleurodesis Patients will then undergo standard medical thoracoscopy in the endoscopy center including the use of moderate sedation, prophylactic antibiotics for 1 week and 20F chest tube insertion at the end of the procedure.
  Interventions: Procedure: Thoracoscopy
- 2 (Experimental): Combined thoracoscopy with pleurodesis and pleurx catheter. In the combined procedure group, a PleurxTM tunnelled catheter will be inserted under ultrasound guidance. As this procedure will be done concurrently with thoracoscopy, there is no estimated increase in endoscopy time.
  Interventions: Other: Thoracoscopy and Pleurx

INTERVENTIONS:
Other: Thoracoscopy and Pleurx — Talc poudrage and tunneled pleural catheter
  Other Names: Pleuroscopy
  Arms: 2
Procedure: Thoracoscopy — Talc poudrage
  Other Names: Pleuroscopy
  Arms: 1

SUMMARY:
Background:

Malignant pleural effusions form a significant proportion of respiratory and oncology work-load. The efficacy of thoracoscopic talc poudrage which is the current standard of care is limited by lung entrapment which prevents lung re-expansion. Thoracoscopy patients also have significant hospital length of stay because chest tube drainage must continue until the pleural space is dry to effect successful pleurodesis.

Alternative management strategies such as tunnelled pleural catheters (bedside ultrasound-guided) enable outpatient management of pleural effusions but have limited pleurodesis rates and do not offer any chance of getting pleural biopsies.

A prospective randomized controlled trial with two arms i.e. thoracoscopic poudrage alone (standard care) versus combined thoracoscopic poudrage and tunnelled pleural catheters. The tunnelled catheters will be inserted at the time of thoracoscopy in the endoscopy centre under ultrasound guidance. The trial is aimed to be completed within 3 years. Primary end-points will be pleurodesis success. The secondary end-points are hospital length-of-stay, complication rates, analgesia requirements, pain scores and quality-of-life scores. Based on power calculations, we aim to recruit 120 patients in each arm.

DETAILED DESCRIPTION:
Malignant effusions are the 2nd commonest cause of exudative effusions and 75% are due to lung, breast and lymphoma primaries. It is estimated that effusions take up about 20% of pulmonologists' work. About 15% of lung cancers have effusions at presentation and 50% will develop effusions during the course of the illness.

The current standard care of a symptomatic malignant effusion is to perform medical thoracoscopy and talc poudrage pleurodesis to prevent recurrence. Reported pleurodesis success with this technique is about 78%. However, this success rate is limited by the presence of lung entrapment that prevents lung re-expansion and effective pleurodesis. Lung entrapment occurs when there is a visceral pleural tumour peel encasing the lungs or when endobronchial tumour causes lung/lobar collapse. Thoracoscopic pleurodesis also results in significant hospital length of stay as chest tubes must stay in situ until the pleural space is dry.

There is also established data on the use of outpatient tunnelled pleural catheters in malignant effusions. Besides providing effective drainage in cases with entrapped lungs, these catheters also result in spontaneous pleurodesis in 42 to 70% of cases. The attraction of the catheters is that it enables early discharge of patients who already have a terminal illness and an extremely poor prognosis (Prognosis is usually about 3-8 months depending on the primary) However, the pleural catheters do not allow biopsies to be taken from the pleura and the pleurodesis rate is both lower and slower than with talc poudrage.

This project hopes to capitalize on the strengths of both methods ie. talc poudrage via thoracoscopy and indwelling pleural catheters, to increase the success of pleurodesis and to decrease hospital stay. Indwelling catheters may improve the success data by draining effusions associated with entrapped lungs that do not usually achieve pleurodesis with talc poudrage alone. These catheters can be left in patients on a long term basis i.e. > 6 months. The attraction of the PleurxTM tunnelled catheter system is the low risk of infections, air leaks (because of a one-way valve) and slippage.4-5 This type of study involving combining both modalities has never been reported in the literature. There is no such trial registered under clinicaltrials.gov. Pilot data (<20 patients) has been previously presented at the American College of Chest Physicians Conference 2006 from Harvard University with promising results.

Current data from our thoracoscopy service in SGH (Jan 2004 to June 2007), shows that our pleurodesis success rate is 78.2%. However, complete success was achieved in 38.1%.7 This data is in keeping with the reported literature and the failures/incomplete successes are attributed to lung entrapment.3 Our data for hospital length of stay is 9.0 ± 4.0 (range 4 to 21) days.

We hypothesized that by combining thoracoscopic talc poudrage with tunnelled catheters, the pleurodesis success rate could be improved by 15% to 93%, complete success to >75 % and hospital length of stay approximately halved to 5 days or less. To test this hypothesis, we want to conduct a prospective, randomized controlled trial comparing thoracoscopic talc poudrage (standard care) to combined talc poudrage with tunnelled pleural catheters.

Procedure:

Patients who meet inclusion/exclusion criteria will be screened by investigators and trial coordinators. After informed consent has been taken, patients will be randomized to either of the study arms. Randomization will be done through a computer generated random list. Baseline data and quality of life scores will be computed.

Patients will then undergo standard medical thoracoscopy in the endoscopy center including the use of moderate sedation, prophylactic antibiotics for 1 week and 20F chest tube insertion at the end of the procedure. The standard of 4-6 g of sterilized talc will be used for talc poudrage.

In the combined procedure group, a PleurxTM tunnelled catheter will be inserted under ultrasound guidance. As this procedure will be done concurrently with thoracoscopy, there is no estimated increase in endoscopy time. If either group of patients is found to have no gross evidence of malignancy at the time of thoracoscopy (ie. empyemas or tuberculous pleurisy), then they will be withdrawn from the study and notified appropriately.

Patients in the standard therapy arm will emerge from the procedure with a chest tube while the intervention arm will have both a chest tube and a tunnelled catheter. In the standard therapy arm, the chest tube will be removed when there is no further air leak and when drainage drops to ≤ 150 ml/day. After chest tube removal, the patient is fit for discharge. In the intervention arm, the chest tube is removed when air leak stops. There will be no need to wait for fluid drainage to decrease and theoretically, the patient can go home on day 3 or 4 with the tunnelled pleural catheter.

Patients in the thoracoscopy only arm will be reviewed at 1 week in the outpatient clinic by the investigators for suture removal and then again at 1 month for evaluation of radiological success. This is the current standard practice. Quality of life assessment will be also done at the one month visit by the trial coordinator. Subsequent follow-ups will be with medical oncology as per standard practice including visits at about 3 months, 6 months and 1 year.

Concurrent chemotherapy and radiotherapy will be allowed as per current standard of care. Concurrent therapy is unlikely to impact our results because non-small cell lung cancers which form the majority of our referrals have poor pleural effusion response to treatment. This is the basis of why pleurodesis is the current standard of care. Chemosensitive tumours like small cell lung cancers, ovarian cancers and lymphomas are seldom referred for symptom management of pleural effusions unless they are refractory to chemotherapy. Again, these patients will not be affected by concurrent 2nd/3rd line therapy. The small group of patients who may be affected by simultaneous oncological management are those who have a first time diagnosis of a chemosensitive tumour like small cell lung cancer or those with a sensitive adenocarcinoma who are managed with Epidermal Growth Factor Tyrosine-kinase (EGRF) inhibitors. These patients comprise <5% of our referrals and will have to analyzed separately in subsets to determine their impact on our data. In our pilot review of SGH thoracoscopy data, these cases formed a tiny proportion (1-2 cases) which prevented any meaningful pilot study analysis.

The patients in the intervention combined treatment arm will be reviewed at outpatient clinic either the next day or within 48 hours. They will undergo drainage via the tunnelled catheter. If drainage is less than 150 ml, the PleurxTM catheter will be removed. Otherwise, the patient will be recalled over the next 24-48 hours till such drainage is achieved. If drainage persists for greater than 5 visits, then these patients will be deemed to have an entrapped lung and will need long term pleural catheterization. Subsequent management will be billed to the patient as part of their usual care. In the rare occurrence of a blocked pleural catheter, a fibrinolytic flush (using streptokinase or alteplase) will be used. This will be done using established protocols for management of blocked catheters.

The primary end points will be pleurodesis/pleural catheter success. Complete success is defined in the literature to be no or minimal re-accumulation of pleural fluid at 30 days. Partial success is defined as partial (≤ 50%) re-accumulation of fluid with some resolution of symptoms and the absence of any further therapeutic interventions at 30 days. If any of these conditions are not met then the procedure is deemed to be a failure.

Secondary endpoints are

1. Hospital length of stay. This will be determined primarily by the primary attending physician based on the patient's medical condition. Patients will be considered 'pleurodesis fit for discharge' the day the chest tube is removed. The chest tube will be removed in the absence of pleural space infection or air-leak (i.e. complications) if the effusion drainage drops to ≤ 150 ml/day and if there is lung re-expansion.
2. Complication rates for infections, bleeding, air-leaks/pneumothorax, tumor seeding of the track
3. Pain scores
4. Analgesia/sedation requirements
5. Talc dose required
6. Quality of life analysis using St George's respiratory questionnaire (pre and post), Borg's scale, ECOG and Karnofsky score.
7. Re-admission and repeat procedure rates for complications related to pleurodesis or re-accumulation of fluid. We aim to track the patients for 1 year.

ELIGIBILITY:
Inclusion criteria:

1. Patients aged ≥ 18 with suspected or known symptomatic malignant pleural effusions (i.e. age >60 or smoking history > 20 pack years or moderate effusion >1/3 hemithorax)
2. Ability and willingness to sign informed consent. See Annex 1 for patient information sheet and informed consent form.
3. Absence of contraindications to thoracoscopy and tunnelled pleural catheters
4. Willingness to comply with follow-up i.e. outpatient follow-up at 1 week and at 1 month for standard intervention; and additional every other day drainage in the intervention group (up to 5 times).

Exclusion criteria:

1. Uncorrected coagulopathy with platelet count ≤ 60 and INR ≥ 1.5.
2. Uncontrolled coughing because of risk of lung puncture and air leaks
3. Severe hypoxemia with a PaO2/FiO2 ratio ≤ 200 or hypercapnia with a PaCO2 ≥ 60 mmHg.
4. Unstable cardiovascular status ie. hemodynamic instability requiring inotropes/vasopressors, recent myocardial infarction < 5 days or uncontrolled arrythmias
5. Uncontrolled psychiatric disorders or absence of a significant caregiver both of which will contraindicate sending the patient home with a tunnelled catheter
6. Previous thoracic surgery/intervention to the affected hemothorax which may have obliterated the pleural space
7. Local skin infections that prevent long term catheter placement
8. Morbid obesity which will increase risks associated with moderate sedation in the endoscopy centre
9. Multi-loculated effusions that will not benefit from drainage
10. Suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary end points will be pleurodesis/pleural catheter success. | 30 days

SECONDARY OUTCOMES:
Hospital length of stay | 1 year
Complication rate/analgesia | 1 year
Quality of life | 1 year
Talc dose | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Devanand Anantham, FCCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Sinagpore General Hospital, Singapore, Singapore

REFERENCES:
- [Result] Shaw P, Agarwal R. Pleurodesis for malignant pleural effusions. Cochrane Database Syst Rev. 2004;(1):CD002916. doi: 10.1002/14651858.CD002916.pub2. PMID 14973997
- [Result] Dresler CM, Olak J, Herndon JE 2nd, Richards WG, Scalzetti E, Fleishman SB, Kernstine KH, Demmy T, Jablons DM, Kohman L, Daniel TM, Haasler GB, Sugarbaker DJ; Cooperative Groups Cancer and Leukemia Group B; Eastern Cooperative Oncology Group; North Central Cooperative Oncology Group; Radiation Therapy Oncology Group. Phase III intergroup study of talc poudrage vs talc slurry sclerosis for malignant pleural effusion. Chest. 2005 Mar;127(3):909-15. doi: 10.1378/chest.127.3.909. PMID 15764775
- [Result] Tremblay A, Michaud G. Single-center experience with 250 tunnelled pleural catheter insertions for malignant pleural effusion. Chest. 2006 Feb;129(2):362-368. doi: 10.1378/chest.129.2.362. PMID 16478853
- [Result] Tremblay A, Mason C, Michaud G. Use of tunnelled catheters for malignant pleural effusions in patients fit for pleurodesis. Eur Respir J. 2007 Oct;30(4):759-62. doi: 10.1183/09031936.00164706. Epub 2007 Jun 13. PMID 17567670